CLINICAL TRIAL: NCT01141010
Title: Effect of Perioperative Psychological Interventions on Maternal Outcomes Undergoing Cesarean Delivery
Brief Title: Effect of Psychological Interventions on Maternal Outcomes Undergoing Cesarean
Acronym: PIMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Confidential Enquiry into Maternal and Child Health (Other)
Responsible Party: DongYing Fu, Nanjing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NJFY1021005; 10NJMS067 (Other Grant/Funding Number: Nanjing Municipal Bureau of Health)
Record Dates: First submitted 2010-06-03; First posted 2010-06-10 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Perioperative Psychology
Keywords: Linguistic; Stress response; Corticosteroid; Cesarean section; Anxiety; Depression; Maternal psychosis
MeSH Terms: conditions — Fractures, Stress; Anxiety Disorders; Depression | interventions — Psycholinguistics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Plain language (Sham Comparator): Conventional plain language will be given without any psychological intervention
  Interventions: Other: Language
- Pre-psycho-language (Active Comparator): Prior surgery psychological linguistic intervention
  Interventions: Other: Language
- Intra-psycho-language (Active Comparator): Intraoperative psychological linguistic intervention
  Interventions: Other: Language
- Post-psycho-language (Active Comparator): Postoperative psychological linguistic intervention
  Interventions: Other: Language
- Combined language (Active Comparator): Psychological linguistic intervention will be given in a combination of pre-, intra- and post-operatively
  Interventions: Other: Language

INTERVENTIONS:
Other: Language — Plain language without psychological intervention
  Arms: Plain language
Other: Language — Psychological linguistic intervention will be given
  Other Names: Psycholinguistic
  Arms: Combined language; Intra-psycho-language; Post-psycho-language; Pre-psycho-language

SUMMARY:
Pregnancy induced psychosis is an essential factor that influencing maternal health postpartum. When gravidas, especially nulliparas, facing labor and delivery, they will undoubtedly encounter burden from their own and surrounding facts. Maternal psychosis takes a large part of women's psychological disorders. No matter which way, either spontaneous or surgical, they would choose, many factors influence their psychological state. Cesarean section poses higher risks for women than vaginal delivery. Therefore, how to seek effective methods to alleviate parturients' psychological stress response possesses pivotal clinical implications. Herein the investigators proposed that different linguistic interventions given pre-, intra- or post-operatively would produce different effect on maternal psychology and internal stress level.

ELIGIBILITY:
Inclusion Criteria:

* Chinese gravidas
* Gestational age >=36 wk
* Nulliparas
* Undergoing selective Cesarean section

Exclusion Criteria:

* With recognition problem
* Used or using centrally acting drugs
* With chronic pain
* Refusal participation
* With existed psychiatric disorders
* With history of psychological diseases
* Contraindications for neuraxial anesthesia

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Self anxiety assessment scale (SAS) | One day prior surgery
  Scorings of SAS evaluation by the patient herself

SECONDARY OUTCOMES:
Self depression assessment scale (SDS) | One day prior surgery
  Scorings of SDS by the patient herself
Visual analog scale of pain (VAS pain) | Five min before surgery (-5 min)
  Patient self assessed pain scorings with a 100 mm (0-100) scale
Saliva cortisol level | One day prior surgery
  Saliva cortisol levels will be measured with EIA
Vital signs | One day prior surgery
  Blood pressure, heart rate, respiratory rate, oral temperature
SAS scorings | 15 min intraoperation
  Scorings of SAS by patient herself
SAS scorings | 30 min postoperation
  Scorings of SAS by the patient herself
SDS scoring | 15 min intraoperation
  Scorings of SDS by patient herself
SDS scoring | 30 min postoperation
  Scorings of SDS by patient herself
VAS pain scoring | Immediately of surgery (0 min)
  VAS scorings of pain by a 100 mm scale
VAS pain scoring | 5 min after surgery begin (+5 min)
  Scorings of VAS pain by a 100 mm scale
VAS pain scoring | Immediately at the end of surgery (this time changed individually)
  Scorings of VAS pain by a 100 mm scale
VAS pain scoring | 3 h after surgery
  Scorings of VAS pain by a 100 mm scale
Saliva cortisol level | 15 min intraoperation
  Saliva cortisol level will be measured with EIA
Saliva cortisol level | 30 min postoperation
  Saliva cortisol level will be measured with EIA
Vital signs | 15 min intraoperation
  Blood pressure, heart rate, respiratory rate, oral temperature
Vital signs | 30 min postoperation
  Blood pressure, heart rate, respiratory rate, oral temperature

CONTACTS AND LOCATIONS:
Overall Officials: DongYing Fu, MSc, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China